CLINICAL TRIAL: NCT05744414
Title: Histological Analysis of AlloMend® Acellular Dermal Matrix Used During the Initial Pre Pectoral Placement of Tissue Expanders for Breast Reconstruction and Evaluated at Time of Permanent Breast Implantation
Brief Title: Histological Analysis of AlloMend® Acellular Dermal Matrix Used in Breast Implant Surgeries
Status: Active, not recruiting | Type: Observational
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Other Study IDs: ADM-002
Record Dates: First submitted 2023-02-09; First posted 2023-02-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Implant; Complications, Infection or Inflammation
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At the time of exchange of tissue expanders to permanent breast implant, tissue specimens of AlloMend® Acellular Dermal Matrix and native tissue will be obtained from eligible and consented patients for histological analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, histologic analysis of biopsied tissue obtained from participants who have undergone a pre-pectoral breast reconstruction or augmentation surgery with expander placement and AlloMend® Acellular Dermal Matrix.

AlloMend® Acellular Dermal Matrix graft incorporation with surrounding native soft tissue using histological assays characterizing host cell infiltration, neovascularization, inflammation, and host replacement of ADM collagen will be studied.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the incorporation of AlloMend® Acellular Dermal Matrix with native surrounding tissue by obtaining up to three, 1 cm diameter biopsies per breast. The samples will then be transported to AlloSource Research and Development Labs for slide preparation and histologic analysis.

This study will be performed at one (1) clinical center in the United States.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* AlloMend® Acellular Dermal Matrix used during the initial prepectoral placement of tissue expanders for breast reconstruction;
* Is scheduled or will be scheduled for a procedure to exchange the tissue expander for permanent breast implant;
* Can understand the requirements of the study, has provided written, informed consent, and to comply with the study protocol.

Exclusion Criteria:

* Mentally compromised (e.g., being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease) in a manner that would compromise his or her ability to consent to participate in the clinical study;
* Subjects who, in the opinion of the investigator, would not be able or willing to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age or greater who have undergone a pre-pectoral placement of tissue expanders for breast reconstruction and will have a histological evaluation of the AlloMend® Acellular Dermal Matrix and native tissue at time of permanent breast implantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
AlloMend® Acellular Dermal Matrix graft incorporation when used in a soft tissue application | At expander/implant exchange surgery; typically 1-3 months post expander placement
  The primary endpoint being evaluated in this study is AlloMend® Acellular Dermal Matrix graft incorporation when used in a soft tissue application. The endpoint will be analyzed from biopsied tissue samples taken during the exchange of expander to permanent breast implant using histological assays characterizing host cell infiltration, neovascularization, inflammation, and host replacement of ADM collagen.

SECONDARY OUTCOMES:
Infection rates | Up to 6 months post expander/implant exchange
  Information collected through clinical standard of care
Seroma rates | Up to 6 months post expander/implant exchange
  Information collected through clinical standard of care
Hematoma rates | Up to 6 months post expander/implant exchange
  Information collected through clinical standard of care
Drain outputs and timing of drain removal | Up to 6 months post expander/implant exchange
  Information collected through clinical standard of care
Revision surgeries | Up to 6 months post expander/implant exchange
  Information collected through clinical standard of care

CONTACTS AND LOCATIONS:
Locations (1):
- Janiga MDs Plastic Surgery and Cosmetic Center, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No